CLINICAL TRIAL: NCT05002556
Title: AFU Registry of the Therapeutic Management and Follow-up of Non-Muscle-Invasive Bladder Cancer
Acronym: TVNIM-AFU
Status: Recruiting | Type: Observational
Sponsor: Association Francaise d'Urologie (Other)
Responsible Party: Sponsor
Other Study IDs: Registry TVNIM-AFU
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Non-Muscle-Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The AFU has set itself the task of setting up a register of medical practices in order to define possible improvements in the therapeutic management and follow-up of NMIBC. In order to obtain representative data, all urologists who are members of the AFU may be invited to include their patients.

DETAILED DESCRIPTION:
BACKGROUND Non-muscle infiltrating bladder tumors are a cancerous pathology with an estimated incidence of 13,000 new cases/year in France. ¾ of new cases are diagnosed at a stage where the cancer is of limited extension to the urothelial mucosa and/or its underlying chorion (non-muscle-invasive bladder cancer NMIBC). The management and follow-up of NMIBCs are performed according to the best practice recommendations issued by the Cancer Committee of the French Urology Association. The risk of recurrence at 1 and 5 years for NMIBC has been estimated in clinical trials to be between 15%-61% and 31%-78%, respectively, depending on grade, stage, number, size, frequency of previous recurrence and presence of carcinoma in situ. In this context, patients should have regular endoscopic examinations to ensure the absence of tumor lesions inside their bladder. Urine cytology pathology is recommended for the detection of recurrence of NMIBC. However, the negative predictive value of this examination does not allow it to be substituted for bladder endoscopy, as the risk of not recognizing a bladder tumor, especially of low grade, is too high. To date, no urinary biomarker has been shown to be clinically useful and their use is not recommended for the non-invasive detection of endovesical tumor recurrence.

Urine sampling is recommended prior to bladder endoscopy for follow-up of NMIBC to ensure urine sterility (CBEU) and to perform urine cytology in patients with high-grade NMIBC and/or carcinoma in situ.

The observational study of the clinical validity of the negative and positive predictive values of the biomarkers in a population of patients followed for a bladder tumor previously characterized is able to demonstrate the possibility of postponing the realization of the cystoscopy according to the tumoral characteristics and the treatments received by the patients.

OBJECTIVES The main objective of the research will be to evaluate the diagnostic performance of biomarkers available in France, performed on a urine sample and providing a binary result (positive: probable presence of a tumor recurrence; negative: probable absence of a tumor recurrence) to the result of the bladder endoscopy performed as part of the routine care for the follow-up of NMIBC: determination of the negative and positive predictive values of biomarkers.

The secondary objectives will be to describe the anatomopathological characteristics, the pathological history and the treatments received in the population, as well as analyze demographic and regional disparities in the treatment profiles of these diseases.

MATERIAL AND METHOD When the patient is included in the study, medical data relating to the patient's pathology, including all previous treatments, will be entered into the register, as well as the name and result of the biomarker carried out before the resection (biopsy). At each follow-up endoscopic examination scheduled in the patient's personalized care plan, the investigating urologist will record its date and endoscopic findings (white light bladder fibroscopy). The name and result of the urine test will also be recorded by the urologist. The performance of the test will be evaluated from these data by calculating sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) and by means of an analysis of variance (ANOVA) to explore possible differences within the test by tumor grade and stage, and according to previous endovesical treatments received.

The inclusion target is 8000 patients in France over a 3-year period.

ELIGIBILITY:
Inclusion Criteria:

* Patient being monitored for a non-muscle-invasive bladder tumor and having undergone a urinary molecular test (biomarker) prior to their resection (biopsy) diagnosis or recurrence,
* AND adult (equal to or > 18 years old),
* AND affiliated with a social security scheme in France,
* AND whose monitoring will be carried out at the recruiting center.

Exclusion Criteria:

* Patient being monitored for a non-urothelial bladder tumor
* Patient refusing follow-up
* Opposition to participation in the study
* Adult protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient being monitored for a non-muscle-invasive bladder tumor and having undergone a urinary molecular test (biomarker) prior to their resection (biopsy) diagnosis or recurrence
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-Free Survival | 5 years
  New bladder cancer (Whether NMIBC or MIBC).
Performance of biomarkers | 5 years
  To evaluate the diagnostic performance of urinary biomarkers available in France, and providing a binary result (positive: probable presence of a tumor recurrence; negative: probable absence of a tumor recurrence) correlated to the result of the bladder endoscopy performed as part of the routine care for the follow-up of NMIBC: determination of the negative and positive predictive values of biomarkers.

SECONDARY OUTCOMES:
Progression-Free Survival | 5 years
  New bladder cancer (MIBC).

CONTACTS AND LOCATIONS:
Locations (27):
- France (27):
  - Centre Hospitalier Beauvais Simone Veil, Beauvais
  - CHU Caen, Caen
  - Hôpital Privé de Sévigné, Cesson-Sévigné
  - Clinique des Cèdres, Cornebarrieu
  - CHD Vendée, La Roche-sur-Yon
  - CHU Kremlin Bicêtre (APHP), Le Kremlin-Bicêtre
  - Clinique Bon Secours, Le Puy-en-Velay
  - Hopital Franco-Britannique Cognac Jay, Levallois-Perret
  - Clinique de la Sauvegarde, Lyon
  - Hopital Edouard Heriot, Lyon
  - Hopital Lyon Sud, Lyon
  - Clinique de la Région Mantaise, Mantes-la-Jolie
  - Hôpital privé Européen - Marseille, Marseille
  - Centre Hospitalier Martigues, Martigues
  - Grand Hôpital de l'Est-Francilien, Meaux
  - Clinique Beau Soleil, Montpellier
  - CHU Nimes, Nîmes
  - Hôpital Pitié-Salpêtrière, Paris
  - GHT Novo - CH René Dubos Pontoise, Pontoise
  - Centre Hospitalier Annecy Genevois, Pringy
  - Clinique la Croix du Sud, Quint-Fonsegrives
  - Clinique Mathilde, Rouen
  - Clinique Saint Hilaire, Rouen
  - Clinique Pasteur, Royan
  - Clinique Saint Germain en laye, Saint-Germain-en-Laye
  - Clinique de l'Union, Saint-Jean
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No